CLINICAL TRIAL: NCT07326904
Title: A Multi-Center, Randomized, Open-Label Study to Evaluate Symptom Relief and Safety After Using Fexuprazan 40 Mg Compared to Esomeprazole 40 Mg in Patients With Gastroesophageal Reflux Disease (GERD)
Brief Title: Study Comparing Fexuprazan and Esomeprazole in Patients With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Ari Fahrial Syam, Consultant Gastroenterologist, Department of Internal Medicine, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP1401262001
Record Dates: First submitted 2025-12-17; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gastro Oesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease (GERD); fexuprazan; esomeprazole; Potassium-competitive acid blockers (P-CABs); Proton pump inhibitors (PPIs); Randomized trial
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — fexuprazan; Esomeprazole

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group interventional design. Eligible participants were randomized in a 1:1 ratio to receive either fexuprazan 40 mg or esomeprazole 40 mg. Each participant remained in the assigned treatment group throughout the study duration.
  All participants received their assigned intervention for an initial treatment period of 4 weeks. Participants who did not achieve adequate symptom relief after the initial treatment period continued treatment with the same assigned intervention for an additional 4 weeks, for a maximum treatment duration of 8 weeks. No crossover between treatment groups occurred at any time during the study.
  Efficacy and safety outcomes were evaluated in parallel between the two treatment groups over the course of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fexuprazan 40 mg (Experimental): Participants assigned to this arm received fexuprazan 40 mg, a potassium-competitive acid blocker (P-CAB), administered orally once daily. The initial treatment period was 4 weeks. Participants who did not achieve adequate symptom relief after the initial treatment period continued treatment with fexuprazan 40 mg for an additional 4 weeks, for a maximum treatment duration of 8 weeks. Treatment adherence and safety were monitored throughout the study period according to the protocol.
  Interventions: Drug: Fexuprazan
- Esomeprazole 40 mg (Active Comparator): Participants assigned to this arm received esomeprazole 40 mg, a proton pump inhibitor, administered orally once daily. The initial treatment period was 4 weeks. Participants who did not achieve adequate symptom relief after the initial treatment period continued treatment with esomeprazole 40 mg for an additional 4 weeks, for a maximum treatment duration of 8 weeks. Treatment adherence and safety were monitored throughout the study period according to the protocol.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Fexuprazan — Fexuprazan was administered orally at a dose of 40 mg once daily. Participants received treatment for an initial period of 4 weeks. Participants who did not achieve adequate symptom relief after the initial treatment period continued treatment with fexuprazan for an additional 4 weeks, for a maximum treatment duration of 8 weeks.
  Arms: Fexuprazan 40 mg
Drug: Esomeprazole — Esomeprazole was administered orally at a dose of 40 mg once daily. Participants received treatment for an initial period of 4 weeks. Participants who did not achieve adequate symptom relief after the initial treatment period continued treatment with esomeprazole for an additional 4 weeks, for a maximum treatment duration of 8 weeks.
  Arms: Esomeprazole 40 mg

SUMMARY:
The goal of this clinical trial was to evaluate the effectiveness and safety of fexuprazan 40 mg for relieving symptoms of gastroesophageal reflux disease (GERD) in adults. The study also compared fexuprazan with esomeprazole 40 mg, a commonly used treatment for GERD.

The main questions this study aimed to answer were:

* Did fexuprazan reduce GERD symptoms such as heartburn and acid regurgitation?
* Was fexuprazan safe and well tolerated compared with esomeprazole?

Researchers compared fexuprazan with esomeprazole to determine whether fexuprazan provided similar symptom relief and safety.

Participants in the study:

* Were randomly assigned to receive fexuprazan 40 mg or esomeprazole 40 mg once daily
* Took the study medication for 4 weeks, with treatment extended up to 8 weeks if symptoms did not improve
* Attended scheduled clinic visits for evaluations
* Completed symptom questionnaires and a daily symptom diary
* Were monitored for side effects and overall safety throughout the study

DETAILED DESCRIPTION:
This multicenter, randomized, open-label, active-controlled clinical study was conducted to evaluate the efficacy and safety of fexuprazan 40 mg, a potassium-competitive acid blocker (P-CAB), compared with esomeprazole 40 mg, a proton pump inhibitor (PPI), in adult patients with gastroesophageal reflux disease (GERD).

GERD is a chronic condition characterized by reflux-related symptoms such as heartburn and acid regurgitation, which can significantly impair quality of life. Although PPIs are widely used as first-line therapy, limitations including delayed onset of action and insufficient control of nocturnal symptoms have been reported. Fexuprazan, a novel P-CAB, inhibits gastric acid secretion through reversible and potassium-competitive inhibition of the H⁺/K⁺-ATPase and has demonstrated rapid onset and sustained acid suppression in prior clinical studies.

Eligible participants were randomized in a 1:1 ratio to receive either fexuprazan 40 mg or esomeprazole 40 mg administered orally once daily. The initial treatment period was 4 weeks. Participants who did not achieve adequate symptom relief after the initial treatment period were eligible to continue the assigned treatment for an additional 4 weeks, for a total treatment duration of up to 8 weeks.

Efficacy was assessed primarily through patient-reported symptom evaluation using validated questionnaires and daily symptom diaries. Safety assessments included monitoring of adverse events, vital signs, physical examinations, and laboratory evaluations throughout the study and during follow-up.

The study was conducted in accordance with the principles of the Declaration of Helsinki, International Council for Harmonisation Good Clinical Practice (ICH-GCP), and applicable local regulatory requirements. Written informed consent was obtained from all participants prior to the performance of any study-related procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years at the time of providing written informed consent
* Male or female participants
* History of gastroesophageal reflux disease (GERD) symptoms, including heartburn and/or acid regurgitation
* GERD symptoms confirmed by:

  * GERD-Q score greater than 7, and
  * Heartburn and/or acid regurgitation occurring on more than 3 days within the last 7 days
* Able to understand the study procedures and complete questionnaires and a daily symptom diary
* Willing and able to provide written informed consent

Exclusion Criteria:

Gastrointestinal conditions:

* Diagnosis of inflammatory bowel disease (Crohn's disease, ulcerative colitis), primary esophageal motility disorders, or pancreatitis
* History of gastric or esophageal surgery affecting acid secretion (except appendectomy, cholecystectomy, or endoscopic polypectomy of benign polyps)
* Alarm symptoms suggestive of gastrointestinal malignancy (e.g., severe dysphagia, odynophagia, gastrointestinal bleeding, anemia, unexplained weight loss), unless malignancy was ruled out

Medical history

* Clinically significant hepatic, renal, endocrine, hematologic, oncologic, or urinary system disease
* History of malignancy within the past 5 years (except non-digestive malignancies that were completely treated with no recurrence for ≥5 years)
* History of psychosis, substance abuse, or alcohol abuse
* Known HIV infection, active hepatitis B, or hepatitis C infection (HCV RNA-positive)

Medication and treatment

* Use of prohibited concomitant medications within 2 weeks prior to enrollment or need for continuous prohibited medication during the study, including:

  * Proton pump inhibitors, potassium-competitive acid blockers, H2-receptor antagonists, or other acid-suppressive agents
  * Certain psychotropic drugs, anticholinergic drugs, antispasmodics, systemic steroids, or mucoprotective agents
* Use of another investigational product within 4 weeks prior to study drug administration

Laboratory findings

* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin ≥2 times the upper limit of normal
* Serum creatinine or blood urea nitrogen ≥2 times the upper limit of normal

Reproductive status

* Pregnant or breastfeeding women
* Women of childbearing potential or male participants who were unwilling to use appropriate contraception during the study

Other

* Known hypersensitivity to the investigational product or comparator drug
* Any condition that, in the opinion of the investigator, made the participant unsuitable for study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Symptom Relief at Week 4 (GERD-Q Score <8) | 4 weeks
  Symptom relief was assessed using the Gastroesophageal Reflux Disease Questionnaire (GERD-Q). The primary outcome was defined as the proportion of participants with a GERD-Q total score of less than 8 at Week 4, indicating adequate relief of GERD symptoms. The GERD-Q is a validated, patient-reported questionnaire that evaluates the frequency and severity of reflux-related symptoms, including heartburn and acid regurgitation.

SECONDARY OUTCOMES:
Proportion of Participants With Symptom Relief at Week 8 (GERD-Q Score <8) | 8 weeks
  The proportion of participants who achieved symptom relief at Week 8, defined as a GERD-Q total score of less than 8. This assessment applied only to participants who continued treatment beyond the initial 4-week period.
Time to Complete Symptom Response | Up to 8 weeks
  Time to complete response was defined as the number of days from first dose of study medication to the first occurrence of complete disappearance of heartburn and/or acid regurgitation for seven consecutive days, based on participant diary records.
Proportion of Participants Without Major GERD Symptoms | Up to 8 weeks
  The proportion of participants without major GERD symptoms (heartburn and/or acid regurgitation) during predefined periods, including the first 7 days, 4 weeks, and 8 weeks after initiation of treatment, as recorded in participant diaries.
Proportion of Days Free of Major GERD Symptoms | Up to 8 weeks
  The proportion of days without heartburn and/or acid regurgitation during the first 7 days, 4 weeks, and 8 weeks after treatment initiation, including daytime, nighttime, and combined daytime/nighttime periods, based on participant diary entries.
Change From Baseline in GERD-Q Score | Baseline to up to 8 weeks
  Change from baseline in GERD-Q total score and symptom frequency at Days 7, Week 4, and Week 8, assessing improvement in reflux-related symptoms over time.
Change From Baseline in GERD-Health-Related Quality of Life (GERD-HRQL) | Baseline to up to 8 weeks
  Change from baseline in GERD-HRQL total score at Days 7, Week 4, and Week 8, evaluating treatment effects on health-related quality of life associated with GERD symptoms.

OTHER OUTCOMES:
Proportion of Participants Without Nocturnal GERD Symptoms | Up to 8 weeks
  The proportion of participants who were not awakened from sleep due to heartburn or acid regurgitation during predefined periods after initiation of study treatment, as recorded in participant diaries.
Proportion of Participants With Relief of Chronic Cough | Up to 8 weeks
  The proportion of participants who experienced relief of chronic cough symptoms during predefined periods after initiation of study treatment, based on participant diary assessments.
Proportion of Participants With Relief of Throat Irritation Sensation | Up to 8 weeks
  The proportion of participants who experienced relief of throat irritation or foreign body sensation during predefined periods after initiation of study treatment, as recorded in participant diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Fahrial Syam, MD, PhD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Universitas Indonesia / RSUPN Dr. Cipto Mangunkusumo
Locations (3):
- Indonesia (3):
  - Menteng Mitra Afia Jakarta Hospital, Jakarta Pusat, DKI Jakarta
  - Islam Cempaka Putih Jakarta Hospital, Jakarta Pusat, DKI Jakarta
  - University of Indonesia Hospital, Depok, West Java

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study protocol and informed consent did not include provisions for data sharing beyond the study investigators. In addition, the data contain sensitive participant information, and sharing IPD is restricted to protect participant confidentiality and comply with local regulations and institutional policies.

REFERENCES:
- [Background] Yang AY, Yoo H, Shin W, Lee YS, Lee H, Kim SE, Kim A. Size-reduced fexuprazan 20 mg demonstrated the optimal bioavailability and bioequivalence with the reference formulation. Transl Clin Pharmacol. 2023 Mar;31(1):40-48. doi: 10.12793/tcp.2023.31.e3. Epub 2023 Mar 22. PMID 37034124
- [Background] Laine L, Sharma P, Mulford DJ, Hunt B, Leifke E, Smith N, Howden CW. Pharmacodynamics and Pharmacokinetics of the Potassium-Competitive Acid Blocker Vonoprazan and the Proton Pump Inhibitor Lansoprazole in US Subjects. Am J Gastroenterol. 2022 Jul 1;117(7):1158-1161. doi: 10.14309/ajg.0000000000001735. Epub 2022 Mar 16. PMID 35294415
- [Background] Shin W, Yang AY, Park H, Lee H, Yoo H, Kim A. A Comparative Pharmacokinetic Study of Fexuprazan 10 mg: Demonstrating Bioequivalence with the Reference Formulation and Evaluating Steady State. Pharmaceuticals (Basel). 2023 Aug 11;16(8):1141. doi: 10.3390/ph16081141. PMID 37631056
- [Background] Kim GH, Choi MG, Kim JI, Lee ST, Chun HJ, Lee KL, Choi SC, Jang JY, Lee YC, Kim JG, Kim KB, Shim KN, Sohn CI, Kim SK, Kim SG, Jang JS, Kim N, Jung HY, Park H, Huh KC, Lee KJ, Hong SJ, Baek S, Han JJ, Lee OY. Efficacy and Safety of Fexuprazan in Patients with Acute or Chronic Gastritis. Gut Liver. 2023 Nov 15;17(6):884-893. doi: 10.5009/gnl220457. Epub 2023 Feb 15. PMID 36789577
- [Background] Kim SI, Lee YC, Cha W, Jung AR, Jang JY, Choi JS, Lee DK, Lee HH, Kwon MS, Lee YS, Eun YG. Efficacy and safety of fexuprazan in patients with symptoms and signs of laryngopharyngeal reflux disease: a randomized clinical trial. Eur Arch Otorhinolaryngol. 2024 Nov;281(11):5873-5883. doi: 10.1007/s00405-024-08877-6. Epub 2024 Aug 8. PMID 39115573
- [Background] Zhuang Q, Liao A, He Q, Liu C, Zheng C, Li X, Liu Y, Wang B, Liu S, Zhang Y, Lin R, Chen H, Deng M, Tang Y, He C, Dai W, Tang H, Gong L, Li L, Xu B, Yang C, Zhou B, Su D, Guo Q, Li B, Zhou Y, Wang X, Fei S, Wu H, Wei S, Peng Z, Wang J, Li Y, Wang H, Deng T, Ding S, Li F, Chen M, Xiao Y. The efficacy and safety of fexuprazan in treating erosive esophagitis: a phase III, randomized, double-blind, multicenter study. J Gastroenterol Hepatol. 2024 Apr;39(4):658-666. doi: 10.1111/jgh.16471. Epub 2024 Jan 22. PMID 38251791
- [Background] Kang N, Kang MG, Lee SE, Kang SY, Jo EJ, Lee JH, Kim SH, Bahn JW, Lee BJ, Song WJ. Efficacy and Safety of Fexuprazan Versus Esomeprazole for Gastroesophageal Reflux Disease-Related Chronic Cough: A Randomized, Double-Blind, Active-Controlled Exploratory Trial. Lung. 2025 Apr 29;203(1):59. doi: 10.1007/s00408-025-00815-5. PMID 40299084
- [Background] Won H, Kim E, Chae J, Lee H, Cho JY, Jang IJ, Chung JY, Kim MG, Lee S. Pharmacokinetic interactions between fexuprazan, a potassium-competitive acid blocker, and nonsteroidal anti-inflammatory drugs in healthy males. Clin Transl Sci. 2024 May;17(5):e13798. doi: 10.1111/cts.13798. PMID 38700290
- [Background] Oh J, Yang E, Jang IJ, Lee H, Yoo H, Chung JY, Lee S, Oh J. Pharmacodynamic and Pharmacokinetic Drug Interactions between Fexuprazan, a Novel Potassium-Competitive Inhibitor, and Aspirin, in Healthy Subjects. Pharmaceutics. 2023 Feb 7;15(2):549. doi: 10.3390/pharmaceutics15020549. PMID 36839870
- [Background] Hwang JG, Jeon I, Park SA, Lee A, Yu KS, Jang IJ, Lee S. Pharmacodynamics and pharmacokinetics of DWP14012 (fexuprazan) in healthy subjects with different ethnicities. Aliment Pharmacol Ther. 2020 Dec;52(11-12):1648-1657. doi: 10.1111/apt.16131. Epub 2020 Oct 27. PMID 33111337
- [Background] Sunwoo J, Oh J, Moon SJ, Ji SC, Lee SH, Yu KS, Kim HS, Lee A, Jang IJ. Safety, tolerability, pharmacodynamics and pharmacokinetics of DWP14012, a novel potassium-competitive acid blocker, in healthy male subjects. Aliment Pharmacol Ther. 2018 Jul;48(2):206-218. doi: 10.1111/apt.14818. Epub 2018 Jun 4. PMID 29863280
- [Background] Lee SP, Sung IK, Lee OY, Choi MG, Huh KC, Jang JY, Chun HJ, Kwon JG, Kim GH, Kim N, Rhee PL, Kim SG, Jung HY, Lee JS, Lee YC, Jung HK, Kim JG, Kim SK, Sohn CI. Randomized Multicenter Study to Evaluate the Efficacy and Safety of Fexuprazan According to the Timing of Dosing in Patients With Erosive Esophagitis. J Neurogastroenterol Motil. 2025 Jan 31;31(1):86-94. doi: 10.5056/jnm24032. Epub 2024 Dec 13. PMID 39667898
- [Background] Hafiz RA, Wong C, Paynter S, David M, Peeters G. The Risk of Community-Acquired Enteric Infection in Proton Pump Inhibitor Therapy: Systematic Review and Meta-analysis. Ann Pharmacother. 2018 Jul;52(7):613-622. doi: 10.1177/1060028018760569. Epub 2018 Feb 18. PMID 29457492
- [Background] Strand DS, Kim D, Peura DA. 25 Years of Proton Pump Inhibitors: A Comprehensive Review. Gut Liver. 2017 Jan 15;11(1):27-37. doi: 10.5009/gnl15502. PMID 27840364
- [Background] Rettura F, Bronzini F, Campigotto M, Lambiase C, Pancetti A, Berti G, Marchi S, de Bortoli N, Zerbib F, Savarino E, Bellini M. Refractory Gastroesophageal Reflux Disease: A Management Update. Front Med (Lausanne). 2021 Nov 1;8:765061. doi: 10.3389/fmed.2021.765061. eCollection 2021. PMID 34790683
- [Background] Kim SE, Kim N, Oh S, Kim HM, Park MI, Lee DH, Jung HC. Predictive factors of response to proton pump inhibitors in korean patients with gastroesophageal reflux disease. J Neurogastroenterol Motil. 2015 Jan 1;21(1):69-77. doi: 10.5056/jnm14078. PMID 25537676
- [Background] Weijenborg PW, Cremonini F, Smout AJ, Bredenoord AJ. PPI therapy is equally effective in well-defined non-erosive reflux disease and in reflux esophagitis: a meta-analysis. Neurogastroenterol Motil. 2012 Aug;24(8):747-57, e350. doi: 10.1111/j.1365-2982.2012.01888.x. Epub 2012 Feb 6. PMID 22309489
- [Background] Yadlapati R, Gyawali CP, Pandolfino JE; CGIT GERD Consensus Conference Participants. AGA Clinical Practice Update on the Personalized Approach to the Evaluation and Management of GERD: Expert Review. Clin Gastroenterol Hepatol. 2022 May;20(5):984-994.e1. doi: 10.1016/j.cgh.2022.01.025. Epub 2022 Feb 2. Erratum In: Clin Gastroenterol Hepatol. 2022 Sep;20(9):2156. doi: 10.1016/j.cgh.2022.05.005. PMID 35123084
- [Background] ASGE Standards of Practice Committee; Desai M, Ruan W, Thosani NC, Amaris M, Scott JS, Saeed A, Abu Dayyeh B, Canto MI, Abidi W, Alipour O, Amateau SK, Cosgrove N, Elhanafi SE, Forbes N, Kohli DR, Kwon RS, Fujii-Lau LL, Machicado JD, Marya NB, Ngamruengphong S, Pawa S, Sheth SG, Thiruvengadam NR, Qumseya BJ; ASGE Standards of Practice Committee Chair. American Society for Gastrointestinal Endoscopy guideline on the diagnosis and management of GERD: summary and recommendations. Gastrointest Endosc. 2025 Feb;101(2):267-284. doi: 10.1016/j.gie.2024.10.008. Epub 2024 Dec 17. PMID 39692638
- [Background] Zhang D, Liu S, Li Z, Wang R. Global, regional and national burden of gastroesophageal reflux disease, 1990-2019: update from the GBD 2019 study. Ann Med. 2022 Dec;54(1):1372-1384. doi: 10.1080/07853890.2022.2074535. PMID 35579516
- [Background] Shaqran TM, Ismaeel MM, Alnuaman AA, Al Ahmad FA, Albalawi GA, Almubarak JN, AlHarbi RS, Alaqidi RS, AlAli YA, Alfawaz KS, Daghriri AA. Epidemiology, Causes, and Management of Gastro-esophageal Reflux Disease: A Systematic Review. Cureus. 2023 Oct 21;15(10):e47420. doi: 10.7759/cureus.47420. eCollection 2023 Oct. PMID 38022211
- [Background] Nirwan JS, Hasan SS, Babar ZU, Conway BR, Ghori MU. Global Prevalence and Risk Factors of Gastro-oesophageal Reflux Disease (GORD): Systematic Review with Meta-analysis. Sci Rep. 2020 Apr 2;10(1):5814. doi: 10.1038/s41598-020-62795-1. PMID 32242117
- [Background] Lee KN, Lee OY, Chun HJ, Kim JI, Kim SK, Lee SW, Park KS, Lee KL, Choi SC, Jang JY, Kim GH, Sung IK, Park MI, Kwon JG, Kim N, Kim JJ, Lee ST, Kim HS, Kim KB, Lee YC, Choi MG, Lee JS, Jung HY, Lee KJ, Kim JH, Chung H. Randomized controlled trial to evaluate the efficacy and safety of fexuprazan compared with esomeprazole in erosive esophagitis. World J Gastroenterol. 2022 Nov 28;28(44):6294-6309. doi: 10.3748/wjg.v28.i44.6294. PMID 36504556
- [Background] Maret-Ouda J, Markar SR, Lagergren J. Gastroesophageal Reflux Disease: A Review. JAMA. 2020 Dec 22;324(24):2536-2547. doi: 10.1001/jama.2020.21360. PMID 33351048
- [Background] Eusebi LH, Ratnakumaran R, Yuan Y, Solaymani-Dodaran M, Bazzoli F, Ford AC. Global prevalence of, and risk factors for, gastro-oesophageal reflux symptoms: a meta-analysis. Gut. 2018 Mar;67(3):430-440. doi: 10.1136/gutjnl-2016-313589. Epub 2017 Feb 23. PMID 28232473
- [Background] Hojo M, Nagahara A, Hahm KB, Iwakiri R, Watanabe T, Rani AA, Zhu Q, Chan FKL, Sollano JD, Kamiya T, Yamaguchi S, Motoya S, Fock KM, Fukudo S, Kachintorn U, Suzuki H, Murakami K; The International Gastroenterology Consensus Symposium Study Group. Management of Gastroesophageal Reflux Disease in Asian Countries: Results of a Questionnaire Survey. Digestion. 2020;101(1):66-79. doi: 10.1159/000504749. Epub 2019 Dec 4. PMID 31801133

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT07326904/Prot_SAP_000.pdf